CLINICAL TRIAL: NCT03890068
Title: A Single-arm, Multicentre, Phase II Clinical Trial of Anlotinib Maintenance Treatment After First-line Anthracycline-based Chemotherapy in Advanced Soft Tissue Sarcoma (ALTER-S006)
Brief Title: Anlotinib Maintenance Treatment for Advanced Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xing Zhang, Vice director of department of medical sarcoma and melanoma,Principal Investigator,Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SunYat-senU-anlotinib
Record Dates: First submitted 2019-03-24; First posted 2019-03-26 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib (Experimental): anlotinib for maintenance treatment a dose of 12 mg once daily (day1-14 PO) in 21-day cycles
  Interventions: Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — 48 subjects with advanced soft tissue sarcoma will receive anlotinib at a dose of 12 mg once daily (day1-14 PO) in 21-day cycles until disease progression (defined by RECIST version 1.1) or unacceptable toxicity.
  Other Names: Anlotinib

SUMMARY:
Anlotinib is a multi-target receptor tyrosine kinase inhibitor. It can inhibit the angiogenesis related kinase, such as Vascular Endothelial Growth Factor Receptor (VEGFR), Fibroblast Growth Factor Receptor(FGFR), Platelet-Derived Growth Factor Receptor(PDGFR), and tumor cell proliferation related kinase c-Kit kinase. Anlotinib is an efficient second line therapeutic agent in treatment for metastatic soft tissue sarcoma which has been approved in clinical trials (ALTER-0203). Therefore, this study evaluates the safety and efficacy of anlotinib as maintenance treatment of disease control in advanced soft tissue sarcoma.

DETAILED DESCRIPTION:
48 cases are preliminarily expected to be included. This study evaluating the safety and efficacy of anlotinib as a maintenance treatment after first-line anthracycline-based chemotherapy in advanced soft tissue sarcoma.

All those participants need to sign informed consent forms for data collection and be used for research purpose before inclusion. Participants remained PR/SD after ≥4 cycles of anthracyclines could be enrolled.

48 subjects with advanced soft tissue sarcoma will receive anlotinib at a dose of 12 mg once daily (day1-14 PO) in 21-day cycles until disease progression (defined by RECIST version 1.1) or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form prior to patient entry;
* 18-70 years , regardless of gender；ECOG :0-2;Expected Survival Time: Over 3 months;
* Subjects with pathologically confirmed advanced synovial sarcoma, leiomyosarcoma, liposarcoma, angiosarcoma, etc. (except malignant peripheral nerve sheath tumor, undifferentiated sarcoma, rhabdomyosarcoma, chondrosarcoma, osteosarcoma, dermato- fibrosarcoma protuberans, gastrointestinal stromal tumor, ewing's sarcoma/primitive neuroectodermal tumor, inflammatory myofibroblastic tumor, and malignant mesothelioma);
* Evaluable disease by imaging or physical exam or measurable disease defined as at least one lesion that can be accurately measured according to RECIST version 1.1.
* PR/SD patients after ≥4 cycles anthracyclines treatment .
* Main organs function is normal.(normal main organs function as defined below: Hemoglobin (Hb) ≥ 80g / L, Neutrophils (ANC) ≥ 1.5 × 109 / L, Platelet count (PLT) ≥ 80 × 109 / L, Serum creatinine (Cr) ≤ 1.5 × normal upper limit (ULN) or creatinine clearance (CCr) ≥ 60ml / min, Blood urea nitrogen (BUN) ≤ 2.5 × normal upper limit (ULN); Total bilirubin (TB) ≤ 1.5 × ULN; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN; If accompanied by liver metastases, ALT and AST ≤ 5 × ULN Albumin (ALB) ≥ 25 g/L. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%).)
* The woman patients of childbearing age who must agree to take contraceptive methods (e.g. intrauterine device, contraceptive pill or condom) during the research and within another 6 months after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; The man patients who must agree to take contraceptive methods during the research and within another 6 months after it.

Exclusion Criteria:

* Prior treatment with anlotinib.
* A history of other malignancy ≤ 5 years previous.
* Systemic anti-tumor therapy, including cytotoxic therapy, signal transduction inhibitors, and immunotherapy, is planned for the first 4 weeks prior to enrollment or during the study. Radiation radiotherapy (EF-RT) was performed within 4 weeks prior to enrollment.
* Unmitigated toxic reactions above grade 1 of CTC AE due to any previous treatment, excluding alopecia.
* Symptoms that affect oral medication and can not be controlled through proper treatment. (such as inability to swallow, chronic diarrhoea and intestinal obstruction, etc.)
* With pleural effusion or ascites, cause respiratory syndrome. (> CTC AE grade 2 dyspnea [grade 2 dyspnea refers to shortness of breath during a small amount of activity; affecting instrumental activities of daily life])
* Symptoms of brain metastases cannot be controlled and treated within less than 2 months.
* Thyroid dysfunction after best support treatment.
* With severe and failed to controlled diseases. (including:1)Uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite optimal drug treatment).2)Arrhythmias with grade II and above myocardial ischemia or myocardial infarction, poor control (including corrected QT interval(QTc) men ≥ 450 ms, women ≥ 470 ms) and ≥ 2 congestive heart failure (New York Heart Association ( NYHA) rating).3)Poor control of diabetes (fasting blood glucose > 10mmol / L).4)Active or uncontrolled serious infection (≥ Common Terminology Criteria for Adverse Event(CTC AE) grade 2 infection);5)Patients with active hepatitis B or hepatitis C (hepatitis B: HBsAg-positive and hepatitis B virus(HBV) DNA ≥ 500 IU/mL; hepatitis C: hepatitis C virus(HCV) RNA-positive and abnormal liver function), or active infection requiring antimicrobial treatment (eg Treated with antibacterial drugs, antiviral drugs, antifungal drugs);6)renal insufficiency: urine routine indicates urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0 g;7)Patients with seizures and need treatment.)
* Accepted surgical treatment, incision biopsy or significant traumatic injury within 28 days before grouping.
* The investigator judged that during the follow-up study, the tumor is very likely to invade the important blood vessels and cause fatal hemorrhage, or the formation of tumor thrombosis with large veins (iliac vessels, inferior vena cava, pulmonary veins, superior vena cava)
* Any major unhealed wound, ulcer, or fracture occurred in a patient who had undergone major surgery or trauma within 4 weeks and/or had any bleeding or bleeding episodes which the degree is bigger than CTCAE 3 grade within 4 weeks prior to enrollment.
* Arteriovenous thrombosis events occurred within 6 months.
* History of psychotropic substance abuse who are unable to quit or have a mental disorder.
* Participated in other anti-tumor clinical trials within 4 weeks.
* The investigator believes that there are any conditions that may damage the subject or result in the subject not being able to meet or perform the research request.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Progress free survival for anlotinib maintenance treatment | until Progressive Disease(PD) or death (up to 24 months)
  Progress free survival defined as the time from first dose of anlotinib treatment until the first date of either objective disease progression or death due to any cause. If the subject did not experience disease progression or death, PFS is defined as the period from the treatment start to the date of the last confirmed progression-free.

SECONDARY OUTCOMES:
Overall Survival | From randomization until death (up to 24 months)
  Overall survival is defined as the time until death due to any cause.
Objective Response Rate | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Objective response rate is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.
Disease Control Rate | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
Safety profile | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Adverse events were recorded throughout the treatment period and 21 days after the last dose and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Xu B, Pan Q, Pan H, Li H, Li X, Chen J, Pang D, Zhang B, Weng D, Peng R, Fang M, Zhang X. Anlotinib as a maintenance treatment for advanced soft tissue sarcoma after first-line chemotherapy (ALTER-S006): a multicentre, open-label, single-arm, phase 2 trial. EClinicalMedicine. 2023 Sep 21;64:102240. doi: 10.1016/j.eclinm.2023.102240. eCollection 2023 Oct. PMID 37767191